CLINICAL TRIAL: NCT06174259
Title: Influence of Intermittent Fasting on Locally Advanced Breast Cancer Patients: a Prospective Randomized Controlled Trial
Brief Title: Influence of Intermittent Fasting on Locally Advanced Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, yostena nagy kamel mekhail, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1998DRXVTF
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Breast Cancer; Intermittent Fasting
Keywords: locally advanced breast cancer; HR positive HER2 negative breast cancer; intermittent fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (Experimental): 16/8 intermittent fasting (limiting foods and calorie-containing beverages to a set window of 8 hours per day) around standard neoadjuvant chemotherapy.
  Interventions: Other: intermittent fasting
- regular diet (No Intervention): Regular diet around standard neoadjuvant chemotherapy

INTERVENTIONS:
Other: intermittent fasting — 16/8 intermittent fasting (limiting foods and calorie-containing beverages to a set window of 8 hours per day)
  Arms: Intermittent fasting

SUMMARY:
Breast cancer is the most common cancer type among women in Egypt and world. Preclinical studies show fasting reduces growth factors and modulates nutrient sensing systems, protecting normal cells against chemotherapy. However, cancer cells are not protected due to Differential Stress Resistance (DSR), making them more vulnerable to chemotherapeutics. This study aims to evaluate intermittent fasting impact on neoadjuvant chemotherapy in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with stage II or III (cT1cN+ or ≥T2 any cN, cM0) breast cancer. - Planned to receive standard neoadjuvant chemotherapy.
* Measurable disease (breast and/or lymph nodes).
* WHO performance status 0-2.
* Being overweight (BMI: 25-29.9 kg/m2) or obese (BMI: ≥30 kg/m2).
* Adequate bone marrow function : white blood cells (WBCs) ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function: bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥50 mL/min
* Patients must be accessible for treatment and follow-up

Exclusion Criteria:

* Serious diseases such as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Diabetes Mellitus.
* Pregnancy or lactating
* Any metabolic disorders that may affect gluconeogenesis or adaptation to fasting periods.
* Previous malignancy.
* Using weight loss medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
pathological response rate | 6months
  Assessment of pathological response using the Miller-Payne grading system; it is a grading system from 1-5 with 5 is the best response

SECONDARY OUTCOMES:
The percentage of patients with grade III/IV toxicity | 6 months
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Grade I/II side effects of chemotherapy | 6 months
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Clinical response | 6months
  Radiological before and after the NACT (neoadjuvant chemotherapy) using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
Body composition changes (fat, muscles, water) | 6 months
  using Bioimpedance analysis (BIA) assessment before, 3months and at the end of NACT
Inflammatory response to chemotherapy. | 6 months
  CRP level
Long term efficacy of treatment | 5 years
  (DFS, OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be published after completing the study in peer reviewed journal